CLINICAL TRIAL: NCT05862753
Title: Evaluating Duration and Depth of Anesthesia by Bispectral Index Induced by an Induction Dose of Etomidate.
Brief Title: Duration and Depth of Anesthesia Induced by a Bolus of Etomidate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SRB2021349
Record Dates: First submitted 2022-01-11; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Etomidate 0,2 mg/kg (Experimental): 8 patients recruited, to receive an injection of bolus of Etomidate at dosage 0,2 mg/kg,
  Interventions: Drug: induction by Etomidate bolus
- Etomidate 0,3 mg/kg (Experimental): 10 patients recruited, to receive an injection of bolus of Etomidate at dosage 0,3 mg/kg
  Interventions: Drug: induction by Etomidate bolus

INTERVENTIONS:
Drug: induction by Etomidate bolus — General anesthesia induction by Etomidate bolus with different concentration in either of the two arms. First arm, has the concentration (0,2 mg/kg) commonly used of Etomidate to induce anesthesia. Second arm, has the concentration (0,3 mg/kg) usually proposed in medical literature.

SUMMARY:
Induction of general anesthesia requires to be safe and to ensure a proper level of anesthesia. A proper anesthesia is sufficient to guarantee loss of consciousness and amnesia and without being too depth leading to a electroencephalogram (EEG) with burst suppression. The depth of anesthesia is monitored by the bispectral index analyse of the EEG, this allows to detect any under- or over-dose of anesthesia. The monitoring works with an unknown algorithm (patent), which evaluate the state of consciousness in the patient.

Etomidate and propofol are commonly use to ensure general anesthesia. Actually, really few litterature has objective informations about the monitoring of Etomidate. The few existant are the old ones and has just a clinical evaluation of the depth of anesthesia (loss of consciousness, loss of breathing, loss of palpebral reflex). Except the fact that these clinical evaluations come from the brain stem, and in fact are not reliable to assess the cortical activity which is reduced by etomidate.

Therefore, some anesthetists are fearful that etomidate is not sufficient to ensure a proper anesthesia to intubate the patient.

This interventionnal study has two purpose. Firstly, a survey will be conduct about the habits and beliefs when use of etomidate.

Secondly, a prospective study will be conduct to monitore with the bispectral index the depth and duration of anesthesia with etomidate.

DETAILED DESCRIPTION:
Protocol with randomization in one of the 2 arms (0.2 vs. 0.3 mg / kg of etomidate), blind to the investigators.

The right dosage will be prepared at the same time by a colleague anesthetist who will not participate in the study according to the randomization envelope that we will give to him earlier. To remain blind to this dosage, it will be diluted with physiological serum up to 30 ml.

These following procedures will be carried out in order:

- Preparation by a colleague of the adequate dose of etomidate, reduced to 20 cc with physiological serum.

No premedication with benzodiazepines (xanax).

* Standard monitoring (ECG + NIBP + SpO2)
* Monitoring the depth of anesthesia by bispectral analysis of the electroencephalography (BIS) trace
* Placement of a peripheral venous line (18 or 20 G) at the bend of the elbow (vein of good size to avoid potential discomfort during the injection of etomidate).
* Preoxygenation with a face mask
* Start remifentanil (20 μg / ml) in AIVOC mode with a site-effect concentration (Cet) of 2 μg / ml) and wait for an equilibration.
* Injection of the induction dose of etomidate over 30 seconds.
* After loss of consciousness, curarisation with 0,6 mg/kg (rocuronium).
* Observation period of the depth of anesthesia. Ventilation support by light ventilation with a face mask.
* Special attention will be paid to avoid any interference with the BIS recording (do not move the patient to set it up, do not turn on the heating blanket).

When the BIS rises above 60, the study stops. The anesthesia is then deepened by administration of propofol and is left to the discretion of the anesthesiologist in charge of the room.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, ASA II, schedule for minor or moderate surgery.

Exclusion Criteria:

* Dependance to alcohol, to drugs, morphinique or psychotrop.
* Epilepsia of severe CNS impairement
* Body weight <70% or >130% to ideal body weight.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
time to loss of consciousness | During general anesthesia induction
  Time for loss of consciousness after etomidate administration
time to loss of palpebral reflex | During general anesthesia induction
  Time to loss of palpebral reflex after etomidate administration
Time for BIS decrease < 60 | During general anesthesia induction
  Time for BIS decrease < 60 after etomidate administration
Duration of adequate general anesthesia | During general anesthesia induction
  Time spent with a bis < 60 after etomidate administration

SECONDARY OUTCOMES:
Presence of secondary effect of etomidate, about presence of myoclonia | During first 15 minutes of general anesthesia
  Myoclonia

OTHER OUTCOMES:
Presence of secondary effect of etomidate, about pain during injection | During first 15 minutes of general anesthesia
  Pain

CONTACTS AND LOCATIONS:
Overall Officials: Céline Boudart, MD, Principal Investigator — Erasme University Hospital
Locations (1):
- Erasme UH, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No